CLINICAL TRIAL: NCT04306263
Title: Evaluation of the Effect of a New Infant Formula With Specific Ingredients on the Development of the Immune System and the Gastrointestinal Health of the Infant
Brief Title: Effect of a New Infant Formula With Specific Ingredients
Acronym: EARLY-TOLERA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laboratorios Ordesa (Industry)
Collaborators: Universidad de Granada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EARLY-TOLERA
Record Dates: First submitted 2020-03-02; First posted 2020-03-12 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Infant Growth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Enriched infant formula (Experimental): Infant formula enriched with dairy ingredients: osteopontin, prebiotics (Human milk oligosaccharide, Glucooligosaccharides) and probiotics.
  Interventions: Dietary Supplement: Enriched infant formula
- Standard formula (Active Comparator): Infants receiving a standard infant formula.
  Interventions: Dietary Supplement: Standard formula
- Breastfeeding arm (Active Comparator): Infants exclusively or predominantly breastfed (>75%).
  Interventions: Dietary Supplement: Breastfeeding arm

INTERVENTIONS:
Dietary Supplement: Enriched infant formula — Infant formula enriched with dairy ingredients: osteopontin, prebiotics and probiotics
  Arms: Enriched infant formula
Dietary Supplement: Standard formula — Infants receiving a standard infant formula.
  Arms: Standard formula
Dietary Supplement: Breastfeeding arm — Infants exclusively or predominantly breastfed (>75%).
  Arms: Breastfeeding arm

SUMMARY:
The purpose of this study is to test whether the addition of certain bioactive ingredients to a new infant formula (HMOs, osteopontin and probiotics) can have a favorable impact on the development of the infant's immune system in the first months of life.

DETAILED DESCRIPTION:
Nowadays, almost all commercial infant formulas resemble the "gold standard" of breast milk in terms of composition of essential nutrients, but it is still a challenge to identify and incorporate certain bioactive components capable of replicating those stimuli typical of breast milk that can program growth, infant development and maturation of the immune system.

The purpose of this study is to test whether the addition of certain bioactive ingredients to a new infant formula (HMOs, osteopontin and probiotics) can have a favorable impact on the development of the infant's immune system in the first months of life.

In addition, considering that the quality of feeding at these early ages will program (Early programming) the health and physiology of the child and the future adult, the study wants to obtain evidence of the effects of this new infant formula on the immune system and the development of the child compared to breast milk during the first year of life, hoping that it promotes proper growth, adequate cognitive development and maturation of the immune system as similar as possible to children fed to the mother's breast.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion age from 0 to 2.5 months of age.
* Gestational age >37 weeks and <41 weeks inclusive.
* Appropriate birth weight appropriate for your gestational age (between 10-90 percentiles).
* APGAR score normal birth to 1' and 5' of 7 - 10.
* Umbilical pH ≥ 7.10.
* Availability to continue throughout the study period.
* Written informed consent

Additional Inclusion Criteria for groups 1 and 2:

* Infants who, at the time of recruitment, have already passed the diet with a majority or exclusive formula for medical reasons, by decision of the parents or any other reason agreed with the pediatrician.

Additional Inclusion Criteria for group 3 (breastfeed infants):

* Infants who have been breastfed until the second month with exclusive or majority breastfeeding.
* Infants who are expected to be exclusively or predominantly breastfed up to 6 months.

Exclusion Criteria:

* Simultaneous participation in other clinical trials.
* Infants suffering from gastrointestinal disorders (allergy and/or intolerance to cow's milk protein or lactose).
* Mother's pathology history and during gestation: neurological diseases, metabolic disorders, type 1 diabetes mellitus, chronic disease (hypothyroidism), maternal malnutrition, TORCH syndrome.
* Treatment of the mother's anxiolytics or antidepressants. Other treatments with drugs potentially harmful to neurodevelopment.
* Inability of the parents to follow up the study (medical decision).

Max Age: 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 231 (Estimated)
Dates: Start 2020-03-02 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Register of infections | From baseline to 12 months
  Register of infant infections through patient diaries completed by parents
Register of fever episodes | From baseline to 12 months.
  Presence and duration of the fever and treatments, through diaries completed by parents
Register of diarrhea episodes | From baseline to 12 months.
  Presence and duration of diarrhea, registered in patients dairies.

SECONDARY OUTCOMES:
Immune response evaluation | At 3, 6 and 12 months of age
  registration of Immunoglobulin secreted in saliva
Demographic data | From baseline to 12 months.
  age of the parents, educational level of the parents, habits and lifestyles of the parents, residence and social environment of the infant.
Obstetric background | Baseline
  Relevant obstetric background
Study of the infant microbiota | At 3, 6 and 12 months.
  Stool bacteria count
Assessment of normal growth of the infant | From baseline to 12 months.
  Evolution of Weight (g), Size (cm) to calculate the Body Mass Index.weight and height will be combined to report BMI in kg/m^2
Infant neurodevelopment | At 12 months
  Analysis of eye movements. Eye tracking technologies is using to assess early cognitive development to evaluate attention domain
Infant neurodevelopment 2 | At 2, 3, 4, 6, 9 and 12 months of age.
  ASQ-3 (Ages & Stages Questionnaires®) ASQ-3 is a set of questionnaires about children's development
Infant neurodevelopment 3 | At 2, 3 and 4 months of life.
  General Movements test (GM´s) GM's is using for the neurological assessment during the first months of life and measures a series of gross movements of variable amplitude and speed involving all body parts
Infant neurodevelopment 4 | 6 and 12 months of age
  Bayley´s Scales of Infant Development III (Spanish version BSID III) is using to evaluate psychomotor and mental development .
Infant neurodevelopment 5 | 12 months of age
  MacArthur Communicative Development Inventory (CDI) . This test assesses the normal process of early language acquisition by various manifestations

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Campoy, MD, Principal Investigator — EURISTIKOS Excellence Centre for Paediatric Research
Locations (1):
- Cristina Campoy, Granada, Andalusia, Spain